CLINICAL TRIAL: NCT04815356
Title: Phase I Study of Anti-CD22 Chimeric Receptor T Cells in Patients With Relapsed/Refractory Hairy Cell Leukemia and Variant
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 210019; 21-C-0019
Record Dates: First submitted 2021-03-24; First posted 2021-03-25 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11-06

CONDITIONS: Hairy Cell Leukemia; Hairy Cell Leukemia Variant
Keywords: CD-22 Expressing Tumor; Chimeric Antigen Receptor; Adoptive Immunotherapy
MeSH Terms: conditions — Leukemia, Hairy Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental therapy: Dose Escalation (Experimental): Escalating doses of autologous anti-CD22-CAR T-cells in subjects to determine the MTD
  Interventions: Biological: CD22CART cell infusion
- Experimental therapy: Dose Expansion (Experimental): Autologous anti-CD22-CAR T-cells at the MTD
  Interventions: Biological: CD22CART cell infusion

INTERVENTIONS:
Biological: CD22CART cell infusion — The treatment regimen will consist of lymphodepleting chemotherapy followed by CD22CART infusion: Days -4 to -2: fludarabine 25 mg/m2/dose Day -2: cyclophosphamide 900 mg/m2/dose Day 0: CD22CART infusion (starting at dose level 1 [DL1]: 1 x 105 transduced CAR-T cells/kg) on Day 0 participants will be evaluated for response at Day 28 post-CD22CART infusion.

SUMMARY:
Background:

CAR (Chimeric Antigen Receptor) T cell therapy is a type of cancer treatment in which a person s T cells (a type of immune cell) are changed in a laboratory to recognize and attack cancer cells. Researchers want to see if this treatment can help people with hairy cell leukemia (HCL).

Objective:

To test whether it is safe to give anti-CD22 CAR T cells to people with HCL.

Eligibility:

Adults ages 18 and older with HCL (classic or variant type) who have already had, are unable to receive, or have refused other standard treatments for their cancer.

Design:

Participants will be screened with the following:

Medical history

Physical exam

Blood and urine tests

Biopsy sample

Electrocardiogram

Echocardiogram

Lung function tests

Imaging scans

Some screening tests will be repeated during the study.

Participants may need to have a catheter placed in a large vein.

Participants will have magnetic resonance imaging of the brain.

Participants will have a neurologic evaluation and fill out questionnaires.

Participants will have leukapheresis. Blood will be removed from the participant. A machine will divide whole blood into red cells, plasma, and lymphocytes. The lymphocytes will be collected. The remaining blood will be returned to the participant.

Participants will get infusions of chemotherapy drugs.

Participants will get an infusion of the anti-CD22 CAR T cells. They will stay at the hospital for 14 days. Then they will have visits twice a week for 1 month.

After treatment, participants will be followed closely for 6 months, and then less frequently for at least 5 years. Then they will have long-term follow-up for 15 years.

DETAILED DESCRIPTION:
Background

* Hairy cell leukemia (HCL) is an indolent CD22+ B-cell leukemia comprising 2% of all leukemias. Most cases of HCL respond well to purine analog chemotherapy and harbor BRAF V600E mutation that can be considered for targeted treatment at the time of relapse. However, there are patients with high-risk HCL such as patients with BRAF wild type IGHV4-34 unmutated HCL who respond poorly to chemotherapy and have poor survival.
* HCL variant (HCLv), also brightly CD22+, resembles HCL morphologically but is more aggressive and responds poorly to standard purine analog chemotherapy. Patients have fewer options of targeted treatment partly due to wild type BRAF. We showed that the overall survival in patients progressed after cladribine-rituximab is less than three years.
* Moxetumomab pasudotox-tdfk is an anti-CD22 recombinant immunotoxin which in 2018 was FDA-approved for adult patients with relapsed/refractory HCL. However, there are patients with HCL and HCLv who progress after treatments with standard purine analog chemotherapy and moxetumomab pasudotox-tdfk, and in the case of classic HCL, even after BRAF +/- MEK inhibition. There is still an unmet need for new treatment options for those with relapsed/refractory disease.
* Adoptive cellular therapy with T-cells genetically modified using viral-based vectors to express chimeric antigen receptors (CAR) targeting the CD22 molecule have demonstrated dramatic clinical responses in patients with CD22+ acute lymphoblastic leukemia (ALL) and non-Hodgkin lymphoma (NHL).
* Moxetumomab pasudotox-tdfk proved that CD22 is a potent target for HCL due to its ubiquitous expression in HCL and HCLv, and cellular therapy represents a promising target for those patients that have progressed after other treatments options with chemotherapy, immunotherapy and targeted therapy. This will be the first trial of anti-CD22 CAR T-cell therapy in the treatment of relapsed/refractory HCL and HCLv.

Objectives

* To assess the safety and feasibility of administering escalating doses of autologous anti-CD22-CAR (M971BBz) engineered T-cells in participants with HCL/HCLv following a cyclophosphamide/fludarabine lymphodepletion regimen.
* Explore whether the administration of anti-CD22-CAR engineered T-cells can mediate antitumor effects in HCL/HCLv.

Eligibility

* HCL/HCLv, after prior treatment with, ineligible for, refusal of, or inability to obtain 1) Rituximab given concurrently with or sequentially after purine analog, 2) moxetumomab pasudotox-tdft, and 3) BRAF-inhibition.
* Need for treatment, either 1) absolute neutrophil count (ANC) <1/nL, 2) hemoglobin (Hgb) <10g/dL, 3) Platelets <100/nL, 4) HCL mass with short axis > 2 cm outside or >0.5 cm inside the central nervous system (CNS), 5) HCL/HCLv count >5/nL in blood or >25/mm^3 in cerebrospinal fluid (CSF), 6) HCL/HCLv count doubling time <6 months and increasing lytic or blastic bone lesions, 7) symptomatic splenomegaly.

  ->= 18 years of age.
* CD22 expression must be detected on greater than 80% of the malignant cells by flow cytometry
* No uncontrolled infection, cardiopulmonary dysfunction, or secondary malignancy requiring treatment.
* No chemotherapy, immunotherapy, or radiation therapy less than or equal to 2 weeks prior to apheresis.

Design

* Peripheral blood mononuclear cells (PBMC) will be obtained by leukapheresis, CD3+ cells enriched and cultured in the presence of anti-CD3/-CD28 beads followed by lentiviral vector supernatant containing the anti-CD22 (M971BBz) CAR.
* On Day -5 (cell infusion is Day 0), participants will begin lymphodepleting chemotherapy comprising fludarabine 30 mg/m2 on Days -5, -4, -3, and -2, and cyclophosphamide 500 mg/m2 on days -3 and -2.
* The CD22-CAR T-cells will be infused on Day 0, with up to a 7 day delay if cells are cryopreserved, if needed for resolution of clinical toxicities, to generate adequate cell numbers, or to facilitate scheduling.
* A Phase I cell dose escalation scheme will be performed primarily using 4 dose levels (1 x 10^5; 3 x 10^5, 1 x 10^6, and 3 x 10^6 transduced T-cells/kg.
* After 2 participants are enrolled at dose level 1 without dose limiting toxicity (DLT) or response, subsequent participants will each be enrolled at increasing dose levels until either DLT or complete response (CR) is observed, after which that dose level will be expanded. Once the maximum tolerated dose (or highest level evaluated) is reached, with 0-1 out of 6 having DLT, an additional 4 participants will be enrolled to provide further assessment of DLTs and for determining a preliminary assessment of the efficacy of the therapy in this participant population.
* Participants will be monitored for toxicity, response and T-cell persistence as well as other biologic correlates.
* Participants who achieve inadequate engraftment of transduced T-cells may receive a 2nd dose of CAR T-cells at a same or higher dose level, with the same or lower dose of lymphodepleting chemotherapy, with results not to affect the primary endpoint of the study.
* Accrual ceiling will be set at 27 to allow for a few inevaluable participants and screen failures.

ELIGIBILITY:
* INCLUSION CRITERIA
* Histologically confirmed diagnosis of HCL or HCLv according to morphological and immunophenotypic criteria of WHO classification [WHO, 2008 revised 2016] of lymphoid neoplasm.
* Participants should have any of the following indications for therapy:

  * ANC <1/nL,
  * Hemoglobin <10g/dL,
  * Platelets<100/nL,
  * Symptomatic splenomegaly,
  * HCL mass with short axis > 2 cm outside or >0.5 cm inside the CNS,
  * HCL/HCLv count >5/nL in blood or >25/mm^3 in CSF,
  * HCL/HCLv count doubling time <6 months and increasing lytic or blastic bone lesions

Participants who have eligible blood counts within 4 weeks from the initiation of study will not be considered ineligible if subsequent blood counts prior to enrollment fluctuate and become ineligible up until the time of enrollment.

* HCL/HCLv, after prior treatment with, ineligible for, refusal of, or inability to obtain 1)rituximab given concurrently with or sequentially after purine analog, 2) moxetumomab pasudotox-tdft, and 3) BRAF-inhibition.
* CD22 expression must be detected on greater than 80% of malignant cells by flow cytometry.
* Participants must have measurable or evaluable disease at the time of enrollment, which may include any evidence of disease including minimal residual disease (MRD) detected by flow cytometry or immunohistochemistry.
* Age >=18 years
* ECOG performance <=2 (Karnofsky >=60%, see Appendix A), participants are exempt from this criterion if poor performance status is related to HCL.
* Participants must have adequate organ function as defined below: Participants must have recovered from the acute side effects of their prior therapy, such that eligibility criteria are met. If participants exhibit minor lab abnormalities that are determined to be related to HCL (not therapy-related), then those participants will be allowed to participate

  * Total bilirubin <= 3 ULN, unless consistent with Gilbert s (ratio between total and direct bilirubin > 5)
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <= 3x upper limit of normal (ULN)
  * Alkaline phosphatase < 2.5 ULN
  * Serum creatinine <= 1.5 mg/dL or creatinine clearance >= 60 mL/min/1.73 m^2 for participants with creatinine levels above institutional normal calculated using eGFR or measured
  * Serum albumin > 2 g/dL
* Prothrombin time (PT)/International Normalized Ratio (INR) < 2.5x ULN (if on warfarin, PT/INR < 3.5x ULN; If on any other anticoagulation, PT < 2.5x ULN
* Fibrinogen >= 0.5x lower limit of normal
* Participants with CNS disease are eligible, with exceptions
* Participants with history of allogeneic stem cell transplantation are eligible if at least 100 days post-transplant, if there is no evidence of active graft-versus-host disease (GVHD) and no longer taking immunosuppressive agents for at least 30 days prior to initiation of study intervention.
* Women of childbearing potential (WOCBP) must agree to use effective contraception (barrier, hormonal, intrauterine device [IUD], abstinence, surgical sterilization) at the study entry and up to 12 months after the last dose of combined chemotherapy or 4 months after cells infusion, whichever is later.

Men must agree to use an effective method of contraception (barrier, surgical sterilization, abstinence) at the study entry and up to 4 months after the last dose of study drug.

* Breastfeeding participants must be willing to discontinue breastfeeding from study treatment initiation through 4 months after the last dose of study drug.
* Ability of participant to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA

* Pregnancy
* Systemic chemotherapy, immunotherapy, or radiation therapy <= 2 weeks prior to apheresis with the following exception:

  * Participants receiving steroids may be enrolled, provided there has been no increase in dose for at least 1 week prior to starting apheresis;
  * For radiation therapy: Radiation therapy must have been completed at least 3 weeks prior to enrollment (including CNS radiation), with the exception that there is no time restriction if the volume of bone marrow treated is less than 10% and also the participant has measurable/evaluable disease outside the radiation port.
* Other anti-neoplastic investigational agents, or antibody-based therapies currently or within 2 weeks prior to apheresis
* Participants taking warfarin
* Prior CAR therapy within 30 days prior to apheresis or prior CAR therapy at any time with evidence for persistence of CAR T cells in blood samples (circulating levels of genetically modified cells of >= 5% by flow cytometry)
* Seropositive for human immunodeficiency virus (HIV) antibody. (Participants with HIV are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy in the future should study results indicate effectiveness.)
* Seropositive for hepatitis C virus (HCV) or positive for hepatitis B surface antigen (HbsAG). Participants who convert to negative will not be excluded for history of positive test.
* Uncontrolled, symptomatic, intercurrent illness including but not limited to infection, congestive heart failure, unstable angina pectoris, cardiac arrhythmia, asthma, chronic obstructive pulmonary disease, psychiatric illness, or social situations that would limit compliance with study requirements or in the opinion of the PI would pose an unacceptable risk to the subject
* History of severe, immediate hypersensitivity reaction attributed to compounds of similar chemical or biologic composition to any agents used in study or in the manufacturing of the cells (i.e., gentamicin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2022-05-23 (Actual); Primary Completion 2036-12-01 (Estimated); Study Completion 2036-12-01 (Estimated)

PRIMARY OUTCOMES:
safety and feasibility | end of treatment
  Fraction of participants at each dose level who experience a toxicity along with the grades and types of toxicity and which can successfully manufacture the targeted dose number
antitumor effect | every year for 15 years
  The fraction of participants who experience a CR among the 10 evaluable participants treated at the MTD or highest safe dose

SECONDARY OUTCOMES:
expansion and persistence | every year for 5 years
  Measure expansion and persistence of adoptively-transferred anti-CD22-CAR-transduced T-cells in the blood and, where possible, the bone marrow
MRD negative CR | every year for 15 years
  Fraction of HCL participants who achieve MRD negative CR following treatment with anti-CD22-CAR engineered T-cells
duration of response | every year for 15 years
  The time between the initial response to therapy and subsequent disease progression or relapse
progression free-survival | every year for 15 years
  Duration of time from the start of treatment until time of disease relapse from PR, disease progression, or death, whichever occurs first
event free survival | every year for 15 years
  Duration of time from the start of treatment until time of disease relapse, disease progression, alternative therapy given (such as radiation), or death, whichever occurs first.
overall survival | every year for for 15 years or until death
  Overall survival (OS) will be determined as the time from the start of the CD22CART infusion until death
time to next treatment | every year for 15 years
  Duration of time from the start of administration of anti-CD22-CAR engineered T-cells to next line of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Kreitman, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2021-C-0019.html